CLINICAL TRIAL: NCT04358380
Title: Liver Injury in Hospitalized Patients With COVID-19 in Latin America: Clinical Characteristics and Prognostic Factors
Brief Title: Liver Injury in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, Coordinator, Austral University, Argentina
Other Study IDs: CIE N° P 20-011
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Liver Injury
Keywords: COVID-19; outcome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without Liver Injury: Hospitalized patients with COVID-19 disease who did not develop liver injury
- Patients with Liver Injury: Hospitalized patients with COVID-19 disease who develop liver injury
  Interventions: Other: Liver injury

INTERVENTIONS:
Other: Liver injury — LFTs elevation or liver decompensation
  Groups: Patients with Liver Injury

SUMMARY:
Coronavirus disease was first diagnosed in December 2019, in the city of Wuhan, China. The World Health Organization recently declared coronavirus disease 2019 (COVID-19) as a pandemic. The infection is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). It is a single-stranded RNA virus, which in humans causes mild respiratory symptoms and generally has a good prognosis. However, in a certain group of patients it manifests as severe pneumonia, respiratory distress syndrome, multiple organ dysfunction and death. The factors associated with a worse prognosis are older than 60 years, the presence of diabetes, cardiovascular disease and obesity. According to studies carried out in the Eastern world, the prevalence of liver injury in patients with COVID-19 disease varies between 14% and 53%, being more prevalent in patients with severe symptoms of COVID-19 disease.

It is not really known whether the liver involvement of patients with SARS-CoV-2 infection is secondary to the direct effect of the virus on the liver. One of the mechanisms of action of SARS-CoV-2 is through the binding to the angiotensin-converting enzyme receptor, which is present in cholangiocytes, this could explain its excretion in faeces. However, liver injury could be due to the immune response generated in the body by the virus with systemic inflammatory response syndrome and the release of inflammatory cytokines such as IL6, generating direct cytopathic damage to the liver. On the other hand, it could be the product of hepatotoxic drugs administered during hospitalization, such as antibiotics, antivirals or non-steroidal anti-inflammatory drugs. Liver biopsy described microvacuolar steatosis, and a mild portal and lobular inflammatory infiltrate .

Therefore, the aim this study is to assess the prevalence of liver complications (liver injury, decompensation of cirrhosis) in patients diagnosed with COVID-19 in Latin America. As secondary objectives, the investigators will describe the clinical characteristics of COVID-19 disease and identify risk factors associated with poor prognosis,

DETAILED DESCRIPTION:
Scenario Multicenter study of patients hospitalized with SARS-CoV-2 in different institutions in Latin America and directed by the Coronavirus and Liver interest group of the Latin American Association for the Study of the Liver (ALEH), coordinated by Dr. Marcelo Silva. This project has been presented to ALEH, which has considered it of high interest and will promote its dissemination among partners and related Associations with the aim of obtaining the greatest participation from the centers in the region.

Design Observational cross-sectional study to describe the prevalence of liver disease in patients hospitalized for SARS-CoV-2. The administrative period of the study will be from 04/25/20 to 12/15/20. The enrollment date of the patients will be the date of the diagnosis of SARS-CoV-2 infection and the date of end of follow-up will be the day of hospital discharge, referral to another center or death.

Participating centers will identify patients who meet the selection criteria during the study period. The diagnosis of SARS-CoV-2 can be made at any time during hospitalization. All included patients will be evaluated and treated according to the specific protocol of each institution. The follow-up period will run until the day of hospital discharge or death.

A specific coded form will be prepared for data registration, which will be subsequently downloaded to a computerized database for subsequent analysis. The exposure variables included in the form will be collected by the investigating doctors.

The following study will be performed following international recommendations for observational studies STROBE guidelines

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 17 years
* Patients with diagnosis of SARS-CoV-2 infection
* Hospitalized patients

Exclusion Criteria:

-

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 17 years hospitalized with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver injury in patients with COVID-19 | through study completion, an average of 6 months
  Hospitalized patients with COVD-19 who developed liver injury

SECONDARY OUTCOMES:
Prognostic factors associated with death | through study completion, an average of 6 months
  Factors associated with worse outcome
Clinical characteristics of patients who developed liver injury | through study completion, an average of 6 months
  Description of patients hospitalized with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo O Silva, MD, Principal Investigator — Austral University
Locations (1):
- Universidad Austral, Pilar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] MacLaren G, Fisher D, Brodie D. Preparing for the Most Critically Ill Patients With COVID-19: The Potential Role of Extracorporeal Membrane Oxygenation. JAMA. 2020 Apr 7;323(13):1245-1246. doi: 10.1001/jama.2020.2342. No abstract available. PMID 32074258
- [Background] Fix OK, Hameed B, Fontana RJ, Kwok RM, McGuire BM, Mulligan DC, Pratt DS, Russo MW, Schilsky ML, Verna EC, Loomba R, Cohen DE, Bezerra JA, Reddy KR, Chung RT. Clinical Best Practice Advice for Hepatology and Liver Transplant Providers During the COVID-19 Pandemic: AASLD Expert Panel Consensus Statement. Hepatology. 2020 Jul;72(1):287-304. doi: 10.1002/hep.31281. PMID 32298473
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190
- [Background] Liu W, Tao ZW, Wang L, Yuan ML, Liu K, Zhou L, Wei S, Deng Y, Liu J, Liu HG, Yang M, Hu Y. Analysis of factors associated with disease outcomes in hospitalized patients with 2019 novel coronavirus disease. Chin Med J (Engl). 2020 May 5;133(9):1032-1038. doi: 10.1097/CM9.0000000000000775. PMID 32118640
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Derived] Mendizabal M, Ridruejo E, Pinero F, Anders M, Padilla M, Toro LG, Torre A, Montes P, Urzua A, Gonzalez Ballerga E, Silveyra MD, Michelato D, Diaz J, Peralta M, Pages J, Garcia SR, Gutierrez Lozano I, Macias Y, Cocozzella D, Chavez-Tapia N, Tagle M, Dominguez A, Varon A, Vera Pozo E, Higuera-de la Tijera F, Bustios C, Conte D, Escajadillo N, Gomez AJ, Tenorio L, Castillo Barradas M, Schinoni MI, Bessone F, Contreras F, Nazal L, Sanchez A, Garcia M, Brutti J, Cabrera MC, Miranda-Zazueta G, Rojas G, Cattaneo M, Castro-Narro G, Rubinstein F, Silva MO. Comparison of different prognostic scores for patients with cirrhosis hospitalized with SARS-CoV-2 infection. Ann Hepatol. 2021 Nov-Dec;25:100350. doi: 10.1016/j.aohep.2021.100350. Epub 2021 Apr 14. PMID 33864948
- [Derived] Mendizabal M, Pinero F, Ridruejo E, Anders M, Silveyra MD, Torre A, Montes P, Urzua A, Pages J, Toro LG, Diaz J, Gonzalez Ballerga E, Miranda-Zazueta G, Peralta M, Gutierrez I, Michelato D, Venturelli MG, Varon A, Vera-Pozo E, Tagle M, Garcia M, Tassara A, Brutti J, Ruiz Garcia S, Bustios C, Escajadillo N, Macias Y, Higuera-de la Tijera F, Gomez AJ, Dominguez A, Castillo-Barradas M, Contreras F, Scarpin A, Schinoni MI, Toledo C, Girala M, Mainardi V, Sanchez A, Bessone F, Rubinstein F, Silva MO. Prospective Latin American cohort evaluating outcomes of patients with COVID-19 and abnormal liver tests on admission. Ann Hepatol. 2021 Mar-Apr;21:100298. doi: 10.1016/j.aohep.2020.100298. Epub 2021 Jan 7. PMID 33359234